CLINICAL TRIAL: NCT05001594
Title: The Effects of a Wearable Vibratory Device on Biomechanics, Quality of Life and Serum Biomarkers After an ACL Reconstruction Surgery
Brief Title: Wearable Vibration Effect on Biomechanics and Biomarkers After ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technion, Israel Institute of Technology (Other)
Collaborators: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Arielle Fischer, Assistant Professor, Technion, Israel Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0089-21-RMB
Record Dates: First submitted 2021-07-22; First posted 2021-08-12 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Knee pathology
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care+ Sham device (No Intervention): Each participant will go through the normal rehabilitation process that follows ACL reconstruction+ a sham device used in the same was as the intervention group.
  The sham device will look the same, will gave the same pressure around the leg, but will not vibrate.
- Usual care+ knee vibratory device (Experimental): Each participant will go through the normal rehabilitation process that follows ACL reconstruction. Additionally, each participant will receive the active device that applies non-invasive vibrational stimulation to the leg for two months, and will be asked to wear it during ambulation for at least an hour per day.
  Interventions: Device: Active vibratory knee device
- Normative data (No Intervention): Healthy participants will go through one session of the full protocol (excluding blood tests):
  * Questionnaires (IKDC, TSK, GAD-7).
  * Biomechanical analysis during walking, stair ambulation, and hoping.
  * Quadriceps and Hamstring strength testing

INTERVENTIONS:
Device: Active vibratory knee device — The active, wearable device is placed above and below the knee joint. The device consists of a sensing module to determine specific points in the gait cycle, a processor to analyze signal from the sensor, and a stimulus module to provide vibratory feedback to the subject.
  Arms: Usual care+ knee vibratory device

SUMMARY:
Anterior cruciate ligament (ACL) injuries account for up to 25% of knee injuries, it is estimated that 32,000-400,000 new cases of ACL tears occur in the USA every year.

The Standard care is twofold; a) ACL reconstruction surgery and b) prolonged rehabilitation period (usually no less than 9 months). However, a large amount of patients do not return to their pre-injury activity level, and up to 30% reinjure their ACL in the following two years.

The wearable system consists of two non-invasive bands, above and below the knee that vibrate during the weight bearing phase while walking.

DETAILED DESCRIPTION:
The objective of this study is to investigate the effect of treatment for ACL reconstruction, including vibrational stimulation and pressure, on locomotion tasks (i.e. walking, stair ascending and descending), muscle function, and pain/function.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Males and females
* Aged 18-50
* Scheduled for an ACL reconstruction in Rambam hospital.
* Hebrew language at mother tongue level

Exclusion Criteria:

* Inability to understand the study protocol.
* Known neuropathies, active cancer, previous fractures in the lower limbs, inflammatory arthritis, implanted electronic devices of any kind.
* Allergies to silver or adhesives.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2023-10-07 (Actual)

PRIMARY OUTCOMES:
Lower limb joints range of motion (Degrees) | Pre-surgery
  Measured by Inertial measurement unit system
Lower limb joints range of motion (Degrees) | 2 months post op
  Measured by Inertial measurement unit system
Lower limb joints range of motion (Degrees) | 4 months post op
  Measured by Inertial measurement unit system
Lower limb joints range of motion (Degrees) | 6 months post op
  Measured by Inertial measurement unit system
Knee strength (Newtons) | Pre-surgery
  Non injured knee, quadriceps and hamstring
Knee strength (Newtons) | 14 days post op
  Non injured knee, quadriceps and hamstring
Knee strength (Newtons) | 2 months post op
  Non injured knee, quadriceps and hamstring
Knee strength (Newtons) | 4 months post op
  Non injured knee, quadriceps and hamstring
Knee strength (Newtons) | 6 months post op
  Non injured knee, quadriceps and hamstring
Knee strength (Newtons) | Pre-surgery
  Injured knee, quadriceps and hamstring
Knee strength (Newtons) | 4 months post op
  Injured knee, quadriceps and hamstring
Knee strength (Newtons) | 6 months post op
  Injured knee, quadriceps and hamstring
The International Knee Documentation Committee (IKDC) Subjective Knee Form | Pre-surgery
  The IKDC total score ranges from 0 to 100, where 100 indicates the highest levels of function and lowest levels of symptoms and 0 indicates the lowest level of function or highest level of symptoms.
The International Knee Documentation Committee (IKDC) Subjective Knee Form | 14 days post op
  The IKDC total score ranges from 0 to 100, where 100 indicates the highest levels of function and lowest levels of symptoms and 0 indicates the lowest level of function or highest level of symptoms.
The International Knee Documentation Committee (IKDC) Subjective Knee Form | 2 months post op
  The IKDC total score ranges from 0 to 100, where 100 indicates the highest levels of function and lowest levels of symptoms and 0 indicates the lowest level of function or highest level of symptoms.
The International Knee Documentation Committee (IKDC) Subjective Knee Form | 4 months post op
  The IKDC total score ranges from 0 to 100, where 100 indicates the highest levels of function and lowest levels of symptoms and 0 indicates the lowest level of function or highest level of symptoms.
The International Knee Documentation Committee (IKDC) Subjective Knee Form | 6 months post op
  The IKDC total score ranges from 0 to 100, where 100 indicates the highest levels of function and lowest levels of symptoms and 0 indicates the lowest level of function or highest level of symptoms.
General Anxiety Disorder-7 (GAD-7) | Pre-surgery
  The GAD-7 total score ranges from 0 to 21, where 21 represents high anxiety and 0 indicates no anxiety
General Anxiety Disorder-7 (GAD-7) | 14 days post op
  The GAD-7 total score ranges from 0 to 21, where 21 represents high anxiety and 0 indicates no anxiety
General Anxiety Disorder-7 (GAD-7) | 2 months post op
  The GAD-7 total score ranges from 0 to 21, where 21 represents high anxiety and 0 indicates no anxiety
General Anxiety Disorder-7 (GAD-7) | 4 months post op
  The GAD-7 total score ranges from 0 to 21, where 21 represents high anxiety and 0 indicates no anxiety
General Anxiety Disorder-7 (GAD-7) | 6 months post op
  The GAD-7 total score ranges from 0 to 21, where 21 represents high anxiety and 0 indicates no anxiety
Tampa Scale of Kinesiophobia (TSK) | Pre-surgery
  The TSK total score ranges from 17 to 68, where 68 represents high kinesiophobia and 17 indicates no kinesiophobia
Tampa Scale of Kinesiophobia (TSK) | 14 days post op
  The TSK total score ranges from 17 to 68, where 68 represents high kinesiophobia and 17 indicates no kinesiophobia
Tampa Scale of Kinesiophobia (TSK) | 2 months post op
  The TSK total score ranges from 17 to 68, where 68 represents high kinesiophobia and 17 indicates no kinesiophobia
Tampa Scale of Kinesiophobia (TSK) | 4 months post op
  The TSK total score ranges from 17 to 68, where 68 represents high kinesiophobia and 17 indicates no kinesiophobia
Tampa Scale of Kinesiophobia (TSK) | 6 months post op
  The TSK total score ranges from 17 to 68, where 68 represents high kinesiophobia and 17 indicates no kinesiophobia

SECONDARY OUTCOMES:
Single-leg hop for distance (cm) | 4 months post op
  Functional assessment
Single-leg hop for distance (cm) | 6 months post op
  Functional assessment
Single-leg drop jump (cm) | 4 months post op, 6 months post op
  Functional assessment
Single-leg drop jump (cm) | 6 months post op
  Functional assessment
Serum Biomarkers (ng/mL) | 4 months post op
  30-minute walk on a treadmill. change in concentration before and after the walk
Surface Electromyography (EMG) | Pre-surgery
  Surface EMG assessment of the quadriceps
Surface EMG | 2 months post op
  Surface EMG assessment of the quadriceps
Surface EMG | 4 months post op
  Surface EMG assessment of the quadriceps
Surface EMG | 6 months post op
  Surface EMG assessment of the quadriceps
Surface EMG | Pre-surgery
  Surface EMG assessment of the hamstrings
Surface EMG | 14 days post op
  Surface EMG assessment of the hamstrings
Surface EMG | 2 months post op
  Surface EMG assessment of the hamstrings
Surface EMG | 4 months post op
  Surface EMG assessment of the hamstrings
Surface EMG | 6 months post op
  Surface EMG assessment of the hamstrings

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Fischer, PhD, Principal Investigator — Technion, Israel Institute of Technology; Bezalel Peskin, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided